CLINICAL TRIAL: NCT02495974
Title: A European Prospective Observational Study Assessing the Effectiveness and Outcomes Associated With Enzalutamide Treatment in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: European Observational Study of Enzalutamide in Metastatic Castration Resistant Prostate Cancer (mCRPC)
Acronym: PREMISE
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 9785-MA-1002
Record Dates: First submitted 2015-07-09; First posted 2015-07-13 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: Xtandi; Enzalutamide; Prostate cancer; Metastatic castration resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with mCRPC prescribed enzalutamide: Oral
  Interventions: Drug: enzalutamide

INTERVENTIONS:
Drug: enzalutamide — oral
  Other Names: Xtandi

SUMMARY:
The purpose of this study is to evaluate the effectiveness of enzalutamide in patients with metastatic castration resistant prostate cancer (mCRPC) in the clinical practice setting as measured by time to treatment failure defined as the time from baseline (treatment initiation) to treatment discontinuation of enzalutamide for any reason including disease progression, skeletal related events, treatment toxicity, patient preference, or death.

ELIGIBILITY:
Inclusion Criteria:

* Men with mCRPC who have been prescribed enzalutamide as part of standard clinical practice
* Germany only: Enzalutamide will be prescribed according to the current SmPC (Summary of Product Characteristics)

Exclusion Criteria:

* Patients with the following will be excluded from study participation in France only:

  * Patients who have previously been treated with abiraterone acetate (Zytiga®) after docetaxel chemotherapy.
  * Patients who have previously been treated with cabazitaxel (Jevtana®)
  * Patients who have previously been treated with Xtandi®
  * Patients taking part in an interventional clinical trial

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with metastatic castration resistant prostate cancer prescribed enzalutamide as part of standard clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 1763 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) | up to 18 months
  Time from baseline (treatment initiation) to treatment discontinuation of enzalutamide for any reason including disease progression, skeletal related events, treatment toxicity, patient preference, or death.

SECONDARY OUTCOMES:
Time to prostate specific antigen (PSA) progression | up to 18 months
  Time from initiation of enzalutamide to the date of PSA progression. PSA progression is defined as a PSA rise of greater than or equal to 25% and an absolute increase of greater than or equal to 2 ng/mL.
PSA response | up to 18 months
Time to disease progression | up to 18 months
  Time from initiation of enzalutamide to the date of radiographic progression, PSA progression or clinical progression according to the investigator's assessment.
Overall Survival (France only) | up to 18 months
  Time from initiation of enzalutamide to death or patient survival at the end of the study.
Treatment duration | up to 18 months
Reason for initiation of treatment with enzalutamide | up to 18 months
Reason for enzalutamide discontinuation | up to 18 months
Subsequent anti-neoplastic therapy for mCRPC | up to 18 months
Time to opiate use | up to 18 months
Pain assessed by Brief Pain Inventory Short Form (BPI-SF) | up to 18 months
  The questionnaire is a patient self-rating scale assessing the level of pain, effect of the pain on activities of daily living, and analgesic use.
Quality of life of participants assessed using EQ-5D-5L | up to 18 months
  EuroQol5 dimension 5 level health state utility index - 5L (EQ-5D-5L) is a standardized instrument for use as a measure of health outcome. It is designed for self-completion by respondents comprising the following dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Quality of life of participants assessed using FACT-P | up to 18 months
  Functional Assessment of Cancer Therapy - Prostate (FACT-P) is a self reported instrument designed to assess patient function in physical, social/family, emotional, and functional well-being and further assesses items for prostate-related symptoms.
Number of participants hospitalized | up to 18 months
Number of visits to health care professionals | up to 18 months
Safety assessed by reported adverse events | up to 18 months
Safety assessed by modification of treatment with enzalutamide as a response to adverse events | up to 18 months
Number of Deaths | up to 18 months
  Deaths defined as deaths due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research Physician, Study Director — Astellas Pharma Europe Ltd.
Locations (182):
- Austria (4):
  - Site AT43001, Bregenz
  - Site AT43005, Innsbruck
  - Site AT43006, Linz
  - Site AT43004, Vienna
- Belgium (11):
  - Site BL32003, Bonheiden, Antwerpen
  - Site BL32004, Brasschaat, Antwerpen
  - Site BL32007, Haine-Saint-Paul, Hainaut
  - Site BL32008, Aalst, Oost-Vlaanderen
  - Site BL32009, Ghent, Oost-Vlaanderen
  - Site BL32010, Sint-Niklaas, Oost-Vlaanderen
  - Site BL32013, Leuven, Vlaams Brabant
  - Site BL32005, Kortrijk, West-Vlaanderen
  - Site BL32001, Brussels
  - Site BL32011, Brussels
  - Site BL32012, Hasselt
- Bulgaria (2):
  - Site BG35903, Plovdiv
  - Site BG35901, Sofia
- Czechia (5):
  - Site CZ42004, Brno
  - Site CZ42007, Jihlava
  - Site CZ42003, Nový Jičín
  - Site CZ42001, Prague
  - Site CZ42006, Prague
- Denmark (4):
  - Site DK45003, Aalborg
  - Site DK45004, Aarhus
  - Site DK45002, Copenhagen
  - Site DK45001, Herlev
- France (56):
  - Site FR33015, Colmar, Alsace
  - Site FR33003, Strasbourg, Alsace
  - Site FR33017, Bordeaux, Aquitaine
  - Site FR33051, Bordeaux, Aquitaine
  - Site FR33018, Bordeaux, Aquitaine
  - Site FR33009, Valence, Auvergne-Rhône-Alpes
  - Site FR33022, Clermont-Ferrand, Auvergne
  - Site FR33006, Aix-en-Provence, Bouches-du-Rhône
  - Site FR33027, Marseille, Bouches-du-Rhône
  - Site FR33041, Marseille, Bouches-du-Rhône
  - Site FR33069, Saint-Martin-Boulogne, Boulogne-sur-Mer
  - Site FR33043, Sens, Bourgogne-Franche-Comté
  - Site FR33026, Brest, Brittany Region
  - Site FR33004, Saint-Grégoire, Brittany Region
  - Site FR33025, Vannes, Brittany Region
  - Site FR33010, Reims, Champagne-Ardenne
  - Site FR33067, Dijon, Côte-d'Or
  - Site FR33062, Longjumeau, Essonne
  - Site FR33033, Évreux, Eure
  - Site FR33002, Quimper, Finistère
  - Site FR33040, Toulouse, Haute-Garonne
  - Site FR33049, Gap, Hautes-Alpes
  - Site FR33039, Lille, Hauts-de-France
  - Site FR33042, Suresnes, Hauts-de-Seine
  - Site FR33020, Tours, Indre-et-Loire
  - Site FR33060, Grenoble, Isère
  - Site FR33050, Bézier, Languedoc-Roussillon
  - Site FR33066, Orléans, Loiret
  - Site FR33061, Vandœuvre-lès-Nancy, Lorraine
  - Site FR33065, Agen, Lot-et-Garonne
  - Site FR33019, Angers, Maine-et-Loire
  - Site FR33007, Nancy, Meurthe-et-Moselle
  - Site FR33059, Albi, Midi-Pyrénées
  - Site FR33021, Coudekerque-Branche, Nord
  - Site FR33063, Beauvais, Oise
  - Site FR33016, Saint-Priest-en-Jarez, Pays de la Loire Region
  - Site FR33070, Amiens, Picardie
  - Site FR33044, Saint-Quentin, Picardie
  - Site FR33028, Clermont-Ferrand, Puy-de-Dôme
  - Site FR33035, Bayonne, Pyrénées-Atlantiques
  - Site FR33012, Lyon, Rhône
  - Site FR33030, Lyon, Rhône
  - Site FR33058, Chalon-Sus-Saone, Saône-et-Loire
  - Site FR33008, Amiens, Somme
  - Site FR33032, Amiens, Somme
  - Site FR33014, Créteil, Val-de-Marne
  - Site FR33037, Saint-Mandé, Val-de-Marne
  - Site FR33011, Toulon, Var
  - Site FR33001, Avignon, Vaucluse
  - Site FR33046, Arras
  - Site FR33054, Hyères
  - Site FR33038, La Chaussée-Saint-Victor
  - Site FR33057, Paris
  - Site FR33034, Paris
  - Site FR33029, Paris
  - Site FR33064, Paris
- Germany (12):
  - Site DE49001, Nürtingen, Baden-Wurttemberg
  - Site DE49016, Wiesbaden, Hesse
  - Site DE49003, Lüneburg, Lower Saxony
  - Site DE49011, Soltau, Lower Saxony
  - Site DE49013, Bonn, North Rhine-Westphalia
  - Site DE49012, Chemnitz, Saxony
  - Site DE49009, Bernburg, Saxony-Anhalt
  - Site DE49015, Kiel, Schleswig-Holstein
  - Site DE49005, Cologne
  - Site DE49006, Rostock
  - Site DE49014, Wuppertal
  - Site DE49010, Würselen
- Greece (12):
  - Site GC30001, Kifissia, Attica
  - Site GC30013, Athens
  - Site GC30007, Athens
  - Site GC30005, Athens
  - Site GC30010, Athens
  - Site GC30003, Athens
  - Site GC30004, Ioannina
  - Site GC30006, Ioannina
  - Site GC30012, Larissa
  - Site GC30008, Thessaloniki
  - Site GC30002, Thessaloniki
  - Site GC30011, Thessaloniki
- Hungary (5):
  - Site HU36006, Debrecen, Hajdú-Bihar
  - Site HU36002, Budapest
  - Site HU36001, Budapest
  - Site HU36005, Szeged
  - Site HU36003, Szombathely
- Ireland (4):
  - Site IR35304, Dublin
  - Site IR35302, Dublin
  - Site IR35305, Dublin
  - Site IR35306, Dublin
- Italy (18):
  - Site IT39001, Meldola, Forlì
  - Site IT39010, Lecco, Lombardy
  - Site IT39009, Rozzano, Milano
  - Site IT39002, Aviano, Pordenone
  - Site IT39013, Candiolo, Torino
  - Site IT39011, Mirano, Venezia
  - Site IT39005, Bari
  - Site IT39012, Catania
  - Site IT39006, Florence
  - Site IT39004, Milan
  - Site IT39017, Milan
  - Site IT39003, Modena
  - Site IT39007, Napoli
  - Site IT39018, Novara
  - Site IT39008, Padua
  - Site IT39015, Palermo
  - Site IT39014, Pisa
  - Site IT39016, Reggio Emilia
- Netherlands (9):
  - Site NL31006, Arnhem
  - Site NL31007, Breda
  - Site NL31005, Doetinchem
  - Site NL31008, Helmond
  - Site NL31001, Hilversum
  - Site NL31004, Hoofddorp
  - Site NL31010, Nieuwegein
  - Site NL31003, The Hague
  - Site NL31011, Zwolle
- Site PT35101, Porto, Portugal
- Site SV38501, Ljubljana, Slovenia
- Spain (14):
  - Site ES34007, Zaragoza, Aragon
  - Site ES34012, Zaragoza, Aragon
  - Site ES34008, Guadalajara, Castille-La Mancha
  - Site ES34009, Toledo, Castille-La Mancha
  - Site ES34013, Barcelona, Catalonia
  - Site ES34011, Lleida, Catalonia
  - Site ES34010, Reus, Catalonia
  - Site ES34004, Badajoz, Extremadura
  - Site ES34006, Cáceres, Extremadura
  - Site ES34005, A Coruña, Galicia
  - Site ES34016, Lugo, Galicia
  - Site ES34003, Ourense, Galicia
  - Site ES34001, Santiago de Compostela, Galicia
  - Site ES34017, Vigo, Galicia
- United Kingdom (24):
  - Site GB44001, Aberdeen, Aberdeenshire
  - Site GB44012, Torquay, Devon
  - Site GB44025, Poole, Dorset
  - Site GB44026, Blackburn, Lancashire
  - Site GB44011, Preston, Lancashire
  - Site GB44004, Boston, Lincolnshire
  - Site GB44002, Lincoln, Lincolnshire
  - Site GB44008, Berkshire, Slough
  - Site GB44013, Weston-super-Mare, Somerset
  - Site GB44007, Treliske, Truro
  - Site GB44009, Swindon, Wiltshire
  - Site GB44005, Worcester, Worcestershire
  - Site GB44023, Birmingham
  - Site GB44010, Brighton
  - Site GB44016, Derby
  - Site GB44020, Guildford
  - Site GB44022, Inverness-shire
  - Site GB44024, Leicester
  - Site GB44003, London
  - Site GB44017, Newcastle upon Tyne
  - Site GB44015, Norfolk
  - Site GB44006, Reading
  - Site GB44014, Taunton
  - Site GB44018, Wolverhampton

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.